CLINICAL TRIAL: NCT04345991
Title: Cohort Multiple Randomized Controlled Trials Open-label of Immune Modulatory Drugs and Other Treatments in COVID-19 Patients - CORIMUNO-CORIPLASM : EFFICACY OF CONVALESCENT PLASMA TO TREAT SARS-COV2 INFECTED PATIENTS
Brief Title: Efficacy of Convalescent Plasma to Treat COVID-19 Patients, a Nested Trial in the CORIMUNO-19 Cohort
Acronym: CORIPLASM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Etablissement Français du Sang (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP200375-10; 2020-001246-18 (EudraCT Number)
Record Dates: First submitted 2020-04-10; First posted 2020-04-15 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Covid19
Keywords: COVID 19; Convalescent plasma
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVID-19 convalescent plasma (Experimental): A plasma unit provided by a COVID-19 convalescent pathogen-reduced plasma will be used for the treatment of the patients.
  Interventions: Drug: Transfusion of COVID-19 convalescent plasma
- Control patients (No Intervention): Control patients will receive the best standard of care

INTERVENTIONS:
Drug: Transfusion of COVID-19 convalescent plasma — Two convalescent plasma units of 200 to 220 ml each will be transfused i.v. as early as possible and no later than 10 days after onset of clinical symptoms. In the absence of acute unforeseen adverse events in the first 3 patients, an additional 2 plasma units of 200/220 ml each will be transfused 24 hours after first 2 units: a total of 4 units / patient
  Arms: COVID-19 convalescent plasma

SUMMARY:
The coronavirus disease 2019 (COVID-19) viral pneumonia is now a worldwide pandemic caused by the Severe acute respiratory virus coronavirus 2 (SARS-CoV-2). The number of cases, and associated mortality has increased dramatically since the first cases in Wuhan, China in December 2019 . To date, no specific treatment has been proven to be effective for COVID-19. Treatment is currently mainly supportive, with in particular mechanical ventilation for the critically ill patients (6.1% in a series of 1099 cases in China). Novel therapeutic approaches are in acute need. In this context, the therapeutic potential associated with convalescent plasma needs to be explored.

The objective of COVIPLASM trial (a nested trial in the CORIMUNO-19 COHORT) is to study the efficacy of convalescent plasma to treat SARS-COV2 infected patients.

DETAILED DESCRIPTION:
Hypothesize: early administration of convalescent plasma containing polyclonal neutralizing Abs may inhibit viral entry and replication (as recently suggested in vitro) and consequently blunt an early pro-inflammatory pathogenic endogenous Ab response.

Potential donors of convalescent plasma will be identified through various means, including hospitals taking care of such patient, practitioners treating outpatients or specific social messaging. Convalescent patients at least 14 to 28 days (per at date regulation regarding blood donation) after the symptoms resolution will be invited to undergo plasma apheresis, pending general eligibility such as an age between 18 and 65 years old and weight not less than 50 kg.

Two convalescent plasma units of 200 to 220 ml each will be transfused i.v. as early as possible and no later than 10 days after onset of clinical symptoms. In the absence of acute unforeseen adverse events in the first 3 patients, an additional 2 plasma units of 200/220 ml each will be transfused 24 hours after first 2 units: a total of 4 units / patient. Transfusion monitoring, treatment and reporting of adverse events will be performed per ANSM hemovigilance regulation regarding transfusion of labile blood products as well as through the specific clinical trial vigilance.

An average of 120 participants will be expected (60 participants in each arm). Availability of ABO compatible plasma will be checked by investigator when a Corimmuno patients is eligible. If so, randomization will be undertaken and patient will be offered to participate in this nested trial if he is allocated to the experimental arm.

An interim analysis is performed at mid-trial, but inclusions are not frozen to wait for the interim analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in the CORIMUNO-19 cohort
* Onset of COVID19 functional signs <8 days (plasma transfusion may occur up to day 10 of onset)
* Mild severity as described in the WHO scale

Exclusion Criteria:

* Pregnancy
* Current documented and uncontrolled bacterial infection.
* Prior severe (grade 3) allergic reactions to plasma transfusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
Survival without needs of ventilator utilization or use of immunomodulatory drugs (other than steroids) | At day 14 after randomization
  Survival without needs of ventilator utilization (including non- invasive ventilation, NIV) or use of immunomodulatory drugs at day 14 of randomization (WHO score < 6) or additional immunomodulatory treatment (other than steroids). Thus, events considered are the need of ventilator use (including non invasive ventilation, NIV, or use of immunomodulatory drugs), or death.
WHO progression scale ≥6 | at day 4 of randomization
  WHO progression scale ≥6 at day 4 of randomization

SECONDARY OUTCOMES:
Severe adverse events | up to 28 days
  Occurrence of severe adverse events known to be associated with plasma transfusion such as transfusion associated circulatory overload (TACO), transfusion related acute lung injury (TRALI), and severe allergy will be reported.
  Occurrence of systemic and/or local (lungs) inflammation associated with convalescent plasma transfusion will also be reported.
WHO progression scale | at 4, 7 and 14 days after randomization
  WHO progression scale at 4, 7 and 14 days after randomization (from stage 4-5 to stage 6 to 10) Uninfected; non viral RNA detected: 0 Asymptomatic; viral RNA detected: 1 Symptomatic; Independent: 2 Symptomatic; Assistance needed: 3 Hospitalized; No oxygen therapy: 4 Hospitalized; oxygen by mask or nasal prongs: 5 Hospitalized; oxygen by NIV or High flow: 6 Intubation and Mechanical ventilation, pO2/FIO2>=150 OR SpO2/FIO2>=200: 7 Mechanical ventilation, (pO2/FIO2<150 OR SpO2/FIO2<200) OR vasopressors (norepinephrine >0.3 microg/kg/min): 8 Mechanical ventilation, pO2/FIO2<150 AND vasopressors (norepinephrine >0.3 microg/kg/min), OR Dialysis OR ECMO: 9 Dead: 10
Overall survival | at 14 and 28 days after randomization
Time from randomization to discharge | Time until discharge up to 28 days
Time to oxygen supply independency | Time until oxygen supply independency up to 28 days
Survival without needs of ventilator utilization | At day 14 after randomization
  Survival without needs of ventilator utilization (including non- invasive ventilation, NIV) at day 14 of randomization (WHO score < 6). Thus, events considered are the need of ventilator use (including non invasive ventilation, NIV), or death.
Survival without use of immunomodulatory drugs | At day 14 after randomization
  Survival without use of immunomodulatory drugs at day 14 of randomization (WHO score < 6). Thus, events considered are use of immunomodulatory drugs, or death.

CONTACTS AND LOCATIONS:
Overall Officials: Karine LACOMBE, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- SMIT, Saint Antoine hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lacombe K, Hueso T, Porcher R, Mekinian A, Chiarabini T, Georgin-Lavialle S, Ader F, Saison J, Martin-Blondel G, De Castro N, Bonnet F, Cazanave C, Francois A, Morel P, Hermine O, Pourcher V, Michel M, Lescure X, Soussi N, Brun P, Pommeret F, Sellier P, Rousset S, Piroth L, Michot JM, Baron G, de Lamballerie X, Mariette X, Tharaux PL, Resche-Rigon M, Ravaud P, Simon T, Tiberghien P. Use of covid-19 convalescent plasma to treat patients admitted to hospital for covid-19 with or without underlying immunodeficiency: open label, randomised clinical trial. BMJ Med. 2023 Oct 27;2(1):e000427. doi: 10.1136/bmjmed-2022-000427. eCollection 2023. PMID 37920150